CLINICAL TRIAL: NCT04471792
Title: Creatine Monohydrate Use and Muscle Stretching in Peripheral Artery Disease
Brief Title: Creatine Use and Muscle Stretching in Peripheral Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Judy Delp, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1150
Record Dates: First submitted 2020-06-20; First posted 2020-07-15 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Muscle stretch; Creatine Monohydrate
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Creatine; Cellulose

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomized, single-blind research design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Creatine monohydrate (Experimental): Creatine Monohydrate will be given at a 5 day loading period (10g/day) followed by a maintenance phase (5 g/day). The objectives of the current trial are to investigate if creatine supplementation plus muscle stretching improves 6-minute walking distance and muscle oxygenation in patients with peripheral artery disease.
  Interventions: Drug: Creatine monohydrate
- Cellulose (Placebo Comparator): These participants will consume a fiber supplement in place of creatine monohydrate at a matched dose with muscle stretching.
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Drug: Creatine monohydrate — Creatine monohydrate will be used in combination with muscle stretching.
  Arms: Creatine monohydrate
Dietary Supplement: Cellulose — Cellulose will be used in combination with muscle stretching.
  Arms: Cellulose

SUMMARY:
To utilize near-infrared spectroscopy to investigate if the research device, which induces muscle stretching, and creatine loading impact submaximal exercise performance in aged and PAD patients. Near-infrared spectroscopy (NIRS)-derived tissue oxygenation responses will be obtained during device placement (muscle stretch) and during a walking test (i.e., six-minute walk test). Muscle oxygenation at rest and during device placement will be assessed with Magnetic Resonance Imaging. It is hypothesized that the stretching protocol will improve both NIRS-derived tissue oxygenation and magnetic resonance-derived muscle oxygenation and that creatine supplementation will further improve phosphorus metabolite muscle performance. All patients will undergo either 4 weeks of stretch training with- or- without creatine supplementation according to previously defined creatine guidelines.

DETAILED DESCRIPTION:
Lower extremity peripheral artery disease (PAD) has been estimated to impact nearly 8.5 million U.S. adults above the age of 40, significantly increasing the rate of morbidity and mortality with concomitant decreases in quality of life. These patients are often given medical therapy (e.g., statins, antiplatelet, anticoagulants) and are also recommended to begin structured exercise programs. However, the limb ischemia that occurs during physical activity in these patients often limits exercise tolerance. A previous study by Bauer and colleagues showed that impaired muscle metabolism is a major contributor to functional limitations in PAD patients. These data are important in that they show alterations in blood flow and metabolic machinery likely impact exercise tolerance. As such, the development of tolerable countermeasures to improve limb blood flow and muscle energetics may increase adherence to exercise therapy and improve health outcomes in PAD patients. Previous work by the investigators has shown that daily muscle stretching, achieved via 30-minutes of ankle dorsiflexion, significantly improved soleus muscle function and muscle blood flow during exercise in a rat model of aging . In a follow-up study, the investigators have also shown that this model improves vascular function and walking function in PAD patients. As noted above, muscle energetics are delayed in PAD patients, so improving the rest-to-exercise transition with creatine supplementation may help PAD patients sustain exercise longer. The investigators are now testing to see if an added supplement can further improve the effects of muscle stretching in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ankle-brachial index (ABI) of 0.90 or less in either leg or clinical diagnosis by a medical doctor (PAD group only)
2. Stable condition for at least 3 months (PAD group only)

Exclusion Criteria:

1. Habitual exercise or cardiovascular rehabilitation program during the past 3 months
2. Critical limb ischemia
3. Blow or above-knee amputation
4. Leg pain at rest
5. Major surgery or lower extremity revascularization in the last 3 months
6. Major medical illness treatment during the prior 12 months
7. Central neurological disease
8. Limited ankle or knee joint range of motion
9. Requirement of oxygen with activity or exercise
10. Heart failure
11. Atrial fibrillation
12. Wheelchair confinement or inability to walk
13. Cognitive disorder
14. Vasculitis problems including Takayasu's arteritis, Berger's disease, collagen disease or Reynaud's disease
15. Overt cardiovascular disease
16. Metabolic disease
17. Renal disease

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Muller-Delp, Ph.D., Principal Investigator — Professor
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hultman E, Soderlund K, Timmons JA, Cederblad G, Greenhaff PL. Muscle creatine loading in men. J Appl Physiol (1985). 1996 Jul;81(1):232-7. doi: 10.1152/jappl.1996.81.1.232. PMID 8828669
- [Background] Hotta K, Behnke BJ, Arjmandi B, Ghosh P, Chen B, Brooks R, Maraj JJ, Elam ML, Maher P, Kurien D, Churchill A, Sepulveda JL, Kabolowsky MB, Christou DD, Muller-Delp JM. Daily muscle stretching enhances blood flow, endothelial function, capillarity, vascular volume and connectivity in aged skeletal muscle. J Physiol. 2018 May 15;596(10):1903-1917. doi: 10.1113/JP275459. Epub 2018 Apr 5. PMID 29623692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 patients were screened. 3 patients were ineligible due to kidney disease and resting leg pain. Thirty patients met eligibility criteria. 8 patients did not respond to follow up and 9 patients lost interest. 13 patients consented to participate and were randomly assigned to either stretch+creatine or stretch+placebo. Zero healthy control participants were enrolled. Only participants with Peripheral Artery Disease were enrolled and randomized to either stretch+creatine or stretch+placebo."
Pre-assignment Details: All 13 patients that were consented completed baseline testing and randomization to either stretch +creatine or stretch + placebo.
Period: Overall Study
Arm/Group | Creatine Monohydrate | Cellulose
Started | 7 (7 patients were assigned to stretch + creatine) | 6 (6 patient were assigned to stretch + placebo (cellulose).)
Completed | 7 (7 patients completed stretch + creatine.) | 6 (6 patients completed stretch +placebo.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Creatine Monohydrate | Cellulose | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Walking Distance
Description: 6-minute walking test. This test measures the distance (in meters) that a patient can walk in 6 minutes.
Time Frame: Baseline and after 4 weeks of intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Creatine Monohydrate | Cellulose
Number analyzed (Participants) | 7 | 6
meters
  Baseline 6MWT Distance | 375 (84) | 411 (72)
  Post-stretching 6MWT Distance | 405 (65) | 425 (83)
Statistical Analysis 1: Comparison: Creatine Monohydrate vs Cellulose; Test type: Superiority; p = 0.38, ANOVA — P=0.380 comparing creatine vs. placebo; Two-way ANOVA for pre vs. post values and for the difference between creatine vs. placebo

2. Secondary Outcome: Change in Percent Oxygenation/Seconds
Description: Near-infrared spectroscopy (NIRS) will be used to measure changes in oxygen saturation (%) in the gastrocnemius muscle. Measurement will be the rate (slope) of the change in oxygen saturation (StO2) per second. Thus rate of rate in oxygenation (slope) = StO2(%)/s = Δ StO2(%)/s
Time Frame: Baseline and after 4 weeks of intervention
Measure: Mean (Standard Deviation); unit: delta StO2 (%/delta time(s)
Arm/Group | Creatine Monohydrate | Cellulose
Number analyzed (Participants) | 6 | 5
delta StO2 (%/delta time(s)
  Baseline Δ StO2(%)/s | 0.59 (0.12) | 0.59 (0.40)
  Post-stretching Δ StO2(%)/s | 0.64 (0.52) | 0.67 (0.44)
Statistical Analysis 1: Comparison: Creatine Monohydrate vs Cellulose; Test type: Superiority; p = 0.883, ANOVA — p=0.883 when comparing effect of creatine to palcebo on rate/change in reperfusion slope; Two-way ANOVA, pre vs. post differences and creatine vs. placebo differences were examined
Statistical Analysis 2: Comparison: Creatine Monohydrate vs Cellulose; Test type: Superiority; p = 0.883, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Creatine Monohydrate | Cellulose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04471792/Prot_003.pdf
  • Statistical Analysis Plan (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04471792/SAP_004.pdf
  • Informed Consent Form (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04471792/ICF_000.pdf